CLINICAL TRIAL: NCT06119750
Title: 4-Day Primary Irritation Patch Test of MIS Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Next Science TM (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSP-020; DS210120 (Other: TKL Research, Inc)
Record Dates: First submitted 2023-04-17; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Healthy; Irritation/Irritant; Reactions Adverse
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Subjects act as their own control. They each receive all three study treatment via patch application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- MIS Solution (Experimental): device under investigation
  Interventions: Device: NS Solution
- Saline (Placebo Comparator): 0.9%
  Interventions: Other: Normal Saline
- Sodium Lauryl Sulfate (Active Comparator): 20%
  Interventions: Other: SLS

INTERVENTIONS:
Device: NS Solution — This will be administered via skin patch.
  Other Names: Antimicrobial Solution
  Arms: MIS Solution
Other: Normal Saline — This will be administered via skin patch.
  Other Names: Negative Control
  Arms: Saline
Other: SLS — This will be administered via skin patch.
  Other Names: Positive Control
  Arms: Sodium Lauryl Sulfate

SUMMARY:
This is a 7 day primary irritation patch test. This study investigates the irritation potential of Next Science MIS Wound Irrigation Solution under standardized conditions compared with an inert control (normal saline) and a known irritant, 20% sodium dodecyl sulfate (also known as sodium lauryl sulfate [SLS]) solution in deionized water [DI] water) on intact skin of healthy human subjects.

DETAILED DESCRIPTION:
In accordance with ISO 10993-10:2010(E), study products will be delivered via dermal patch at 15 and 30 minutes (min) and up to 1-hour (h), 2-h, 3-h, 4-h and then, pending results, 24-h (evaluated up to at least 48-h) continuous exposure. Response rate will be evaluated immediately after application then 1 h, 2 h, 24 h, 48 h, and then 72 h post-exposure.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible for inclusion in the study were those who:

  1. Were male or female, 18 - 75 years of age, in general good health (confirmed by medical history);
  2. If females of childbearing potential, were using an acceptable form of birth control (i.e., oral contraceptive, intra-uterine device [IUD], diaphragm, condom, abstinence, bilateral tubal ligation, or are in a monogamous relationship with a partner who had a vasectomy);
  3. In the case of females of childbearing potential, had a negative urine pregnancy test (UPT) at Screening (a woman was considered to be of non-childbearing potential if she was postmenopausal for at least 12 months or was surgically sterile [hysterectomy, bilateral oophorectomy]);
  4. Agreed not to use systemic/topical corticosteroids within 3 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
  5. Agreed not to use systemic/topical analgesics such as aspirin (81 mg daily aspirin were allowed at the discretion of the Investigator), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to and during the study (occasional use of acetaminophen was permitted);
  6. Were free of any systemic or dermatologic disorder which, in the opinion of the investigative personnel, interfered with the study results or increased the risk of adverse events (AEs);
  7. Were of any skin type or race providing the skin pigmentation allowed for discernment of erythema;
  8. Completed a medical screening procedure; and
  9. Read, understood, and signed an informed consent agreement

Exclusion Criteria:

* Had any visible skin disease at the study site which, in the opinion of the investigative personnel, would have interfered with the evaluation; 2. Were receiving systematic or topical drugs or medication which, in the opinion of the investigative personnel, would have interfered with the study results; 3. Had psoriasis and/or active atopic dermatitis/eczema; and/or 4. Had a known sensitivity to cosmetics, skin care products, or topical drugs as related to the material being evaluated. 5. Had a history of allergies or sensitivity to study material being tested. 6. Were pregnant women. 7. Were women who were breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — at least 1/3 males and 1/3 females
Enrollment: 33 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of wound solution on healthy volunteers when applied to the skin. | 7 days
  Response Grade of Irritation